CLINICAL TRIAL: NCT06412471
Title: A Phase II Study of SSGJ-707 Combination Therapy in Advanced NSCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-707-NSCLC-II-02
Record Dates: First submitted 2024-04-26; First posted 2024-05-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-05

CONDITIONS: First-line Advanced NSCLC Patients
MeSH Terms: interventions — Carboplatin; Pemetrexed; Paclitaxel; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm 1 (Experimental): dose level 1 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: Pemetrexed
- Arm 2 (Experimental): dose level 2 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: Pemetrexed
- Arm 3 (Experimental): dose level 3 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: Pemetrexed
- Arm 4 (Experimental): PD-1/L1 combined with chemotherapy
  Interventions: Drug: carboplatin; Drug: Pemetrexed; Drug: PD-1/L1
- Arm 5 (Experimental): dose level 1 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- Arm 6 (Experimental): dose level 2 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- Arm 7 (Experimental): dose level 3 of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- Arm 8 (Experimental): Selected dose of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- Arm 9 (Experimental): Selected dose of SSGJ-707 combined with chemotherapy
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: Paclitaxel-albumin
- Arm 10 (Experimental): PD-1/L1 combined with chemotherapy
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: PD-1/L1

INTERVENTIONS:
Drug: SSGJ-707 — bispecific antibody
  Arms: Arm 1; Arm 2; Arm 3; Arm 5; Arm 6; Arm 7; Arm 8; Arm 9
Drug: carboplatin — chemotherapy
Drug: Pemetrexed — chemotherapy
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: paclitaxel — chemotherapy
  Arms: Arm 10; Arm 5; Arm 6; Arm 7; Arm 8
Drug: PD-1/L1 — Immune checkpoint inhibitors
  Arms: Arm 10; Arm 4
Drug: Paclitaxel-albumin — chemotherapy
  Arms: Arm 9

SUMMARY:
This study includes two parts, part A is for non-squamous NSCLC and part B is for squamous NSCLC.

DETAILED DESCRIPTION:
This study is a study of SSGJ-707 combination therapy in First-line advanced NSCLC Patients. This study includes two parts, part A is for non-squamous NSCLC and part B is for squamous NSCLC. Each part will assess the efficacy and safety of the preset several dose levels of SSGJ-707 in advanced NSCLC Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or metastatic NSCLC .
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=3 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-707 The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  Objective response rate
Safety and tolerability | 12 months
  Safety and tolerability assessed by incidence and severity of adverse events

SECONDARY OUTCOMES:
PFS | 24 months
  The efficacy end points

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of The Hunan Cancer Hospital, Changsha, China

IPD SHARING:
Plan to Share IPD: No